CLINICAL TRIAL: NCT07092696
Title: Induction Immunotherapy Combined With Chemotherapy Followed by Concurrent Chemoradiotherap and Immunotherapy for Advanced Cervical Cancer: An Open-Label, Single-Arm, Phase II Trial
Brief Title: Induction Immunotherapy Combined With Chemotherapy Followed by Concurrent Chemoradiotherap and Immunotherapy for Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250419
Record Dates: First submitted 2025-07-16; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 arm (Experimental): Induction PD-1 inhibitor followed by PD-1 maintenance administered concurrently with chemoradiotherapy and continued after completion.
  Interventions: Drug: Toripalimab; Radiation: Pelvic External-Beam Radiotherapy (EBRT)

INTERVENTIONS:
Drug: Toripalimab — Induction chemo-immunotherapy (platinum-based tri-weekly regimen)
  * Paclitaxel 175 mg/m² IV on day 1
  * Cisplatin 50 mg/m² IV on day 1 or carboplatin AUC 4-5 IV on day 1
  * Toripalimab 240 mg IV on day 1, administered immediately before each chemotherapy infusion Cycle length: every 3 weeks Number of cycles: 2 Concurrent chemoradiotherapy (weekly regimen)
  * Radiation therapy delivered according to institutional protocol
  * Cisplatin 40 mg/m² IV once weekly
  * Toripalimab 240 mg IV on day 1 of every 3-week cycle, given before chemotherapy Cycle length: every 3 weeks during radiotherapy
  Maintenance immunotherapy
  • Toripalimab 240 mg IV on day 1 every 3 weeks (Q3W) Duration: 1 year (total 13 cycles)
Radiation: Pelvic External-Beam Radiotherapy (EBRT) — * PTV: 6 MV photons, 1.80 Gy per fraction × 28 fractions = 50.4 Gy.
  * PGTVnd: 6 MV photons, 2.14 Gy per fraction × 28 fractions = 59.92 Gy. Brachytherapy:Dose prescriptions
  * Dose: 7.00 Gy per fraction × 4 fractions = 28.0 Gy.

SUMMARY:
To explore the efficacy and tolerability of a platinum-based regimen combined with the PD-1 antibody toripalimab administered prior to concurrent chemoradiotherapy in patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
At the 2024 American Society of Clinical Oncology (ASCO) Annual Meeting, investigators reported that neoadjuvant camrelizumab combined with induction chemotherapy, followed by camrelizumab plus concurrent chemoradiotherapy and subsequent camrelizumab maintenance, achieved an overall response rate of 100 % in patients with locally advanced cervical cancer, with an acceptable safety profile.

Pre-clinical studies have suggested that concurrent chemoradiotherapy may dampen immune activation in cervical cancer, including reductions in the CD4+/CD8+ T-cell ratio and decreased T-cell receptor (TCR) diversity. These findings imply that administration of immunotherapy prior to chemoradiotherapy might be more effective than giving it concomitantly or afterwards.

Informed by these clinical and translational data, we propose to conduct an initial, prospective phase II trial to evaluate the efficacy and safety of neoadjuvant chemo-immunotherapy followed by concurrent chemoradiotherapy plus immunotherapy in patients with locally advanced cervical cancer, thereby laying the groundwork for a subsequent phase III investigation.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years.

  * Histologically confirmed, previously untreated locally advanced cervical cancer of squamous, adenocarcinoma, or adenosquamous type.
  * At least one measurable lesion that has not received prior local therapy (non-nodal lesion ≥ 10 mm longest diameter or pathological lymph node ≥ 15 mm short axis, per RECIST 1.1).
  * Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
  * Estimated life expectancy ≥ 6 months.
  * Investigator-assessed eligibility for concurrent chemoradiotherapy.
  * No clinically significant active bleeding.
  * Laboratory values: WBC > 4 × 10⁹/L; platelets > 100 × 10⁹/L.
  * No history of other malignancies.
  * Women of child-bearing potential must have a negative serum pregnancy test and use effective contraception throughout the study.
  * Written informed consent obtained prior to any study-related procedures.

Exclusion Criteria:

* Tumor recurrence or distant metastasis at screening.

  * Active autoimmune disease requiring systemic therapy, or any chronic condition requiring long-term high-dose corticosteroids (≥10 mg/day prednisone or equivalent) or other immunosuppressive agents.
  * Systemic corticosteroids (>10 mg/day prednisone or equivalent) or any other immunosuppressive drugs within 14 days before first study dose or anticipated during the study.
  * Live-attenuated vaccination within 30 days before first dose or planned during the study.
  * Prior organ transplantation or known HIV infection.
  * Active hepatitis B (HBV DNA >2000 IU/mL or >10⁴ copies/mL, or HBsAg positive) or active hepatitis C (HCV RNA >10³ copies/mL); co-infection with both viruses is also excluded.
  * Prior therapy with any agent targeting PD-1, PD-L1, PD-L2, CD137, CTLA-4 (e.g., ipilimumab), or any other antibody or drug that modulates T-cell co-stimulation or checkpoint pathways.
  * Known hypersensitivity to monoclonal antibodies, fusion proteins, or any excipients in the investigational products.
  * History of another malignancy within the past 5 years, except adequately treated cervical carcinoma in situ, basal-cell carcinoma of the skin, or other localized malignancies considered cured.
  * Severe non-surgical comorbidity or acute infection.
  * Peripheral neuropathy > Grade 1 (NCI-CTCAE).
  * Inadequate hematologic or organ function:
  * WBC < 4.0 × 10⁹/L, ANC < 1.5 × 10⁹/L, platelets < 100 × 10⁹/L, Hb < 90 g/L
  * TBIL > 1.5 × ULN, ALT/AST > 2.5 × ULN, BUN > 1.5 × ULN, creatinine > 1.5 × ULN
  * Symptomatic brain metastases.
  * Clinically significant cardiac arrhythmias, myocardial ischemia, severe conduction block, heart failure, or severe valvular disease.
  * Severe bone-marrow failure.
  * Uncontrolled psychiatric illness.
  * Pregnant or lactating women.
  * Investigator-judged unsuitability for the trial.
  * Concurrent participation in another interventional clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1

SECONDARY OUTCOMES:
Disease Free Survival | 3 year
  Time from diagnosis of disease to disease recurrence or death due to any cause
Overall survival | 3 year
  Time from diagnosis of disease of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute&Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No